CLINICAL TRIAL: NCT02218970
Title: The Effect of Muscular Strength Training in Patients With Drug Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/640
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Substance-related Disorders
Keywords: rehabilitation; strength training; muscle strength; physical fitness
MeSH Terms: conditions — Substance-Related Disorders | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- strength training (Experimental): Strength training for leg muscles during10 weeks, 3 times a week: hack squat and plantar flexion, standing upright in a hack squat machine and lying down in a calf rise machine. Exercises will be carried out at 85% of 1-RM intensity under supervision at the institution where participants are having their SUD treatment.
  Interventions: Behavioral: strength training
- control (Other): patients treated for substance-related disorder but not participating in strength training intervention (no training control group)
  Interventions: Behavioral: no training (control)

INTERVENTIONS:
Behavioral: strength training
  Arms: strength training
Behavioral: no training (control)
  Arms: control

SUMMARY:
Physical health does not have a high priority in today's treatment of patients with substance use disorder (SUD). SUD patients have a poor physical health not only due to injuries related to the substance abuse, but also because of the addiction-related lifestyle. There are few studies today that provide information about SUD patient's physical health, and especially there is little information about their muscular strength. One of the project's aims is to measure muscular strength in SUD patients who are being treated for their addiction, and see if they have decreased neuromuscular function. If so, we will investigate the effect of maximal strength training on neuromuscular function in these patients.

ELIGIBILITY:
Inclusion Criteria:

* being treated for drug abuse
* not using drugs during intervention period

Exclusion Criteria:

* participated in strength training in previous 6 months
* cardiovascular disease
* any other disease that impedes to finish tests
* not showing up for testing sessions
* carried out less than 85% of planned exercise sessions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
muscle strength | 10 weeks
  Assessed peripheral muscle strength by one repetition maximum test (1RM)

CONTACTS AND LOCATIONS:
Overall Officials: Grete Flemmen, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Rusbehandling Midt-Norge H, Trondheim, Norway

REFERENCES:
- [Result] Unhjem R, Flemmen G, Hoff J, Wang E. Maximal strength training as physical rehabilitation for patients with substance use disorder; a randomized controlled trial. BMC Sports Sci Med Rehabil. 2016 Mar 31;8:7. doi: 10.1186/s13102-016-0032-2. eCollection 2016. PMID 27042312